CLINICAL TRIAL: NCT04454983
Title: Lipiflow vs iLux Patient Acceptance and Comfort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epstein, Arthur B., OD, FAAO (Individual)
Collaborators: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Arthur Epstein, Director of Dry Eye and Ocular Surface Disease, Epstein, Arthur B., OD, FAAO
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PEC-Sep2019-Lipi-iLux
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye
Keywords: meibomian gland dysfunction; dry eye; Lipiflow; iLux
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: This study is an open-label, single site, crossover trial comparing LipiFlow Thermal Pulsation System to the iLux System based on patient acceptance, comfort, and preference.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lipiflow - All Subjects (Experimental): Both Lipiflow and iLux procedures were performed bilaterally on all subjects on the same day. Subjects were randomized to which procedure they received first. There was a 1-hour wait between procedures.
  Interventions: Device: Lipiflow Thermal Pulsation System
- iLux - All Subjects (Experimental): Both Lipiflow and iLux procedures were performed bilaterally on all subjects on the same day. Subjects were randomized to which procedure they received first. There was a 1-hour wait between procedures.
  Interventions: Device: iLux System

INTERVENTIONS:
Device: Lipiflow Thermal Pulsation System — The LipiFlow Console provides the user interface and control elements of the system, including all software, algorithms and control elements. The Activator, a single-use sterile device, delivers automated therapeutic energies to each meibomian gland. Its contoured design vaults the cornea and protects the eye allowing a maximum therapeutic temperature of 43 degrees Celsius to reach glands from the inner eyelid. Insulation protects the cornea from exceeding a safe 39.5 degrees Celsius, while a pressure feedback loop sends pulsed sequences to expel blockages. Force equalization protects the globe from pressure transmission by focusing energy only on the eyelid. Delivered through the LipiFlow Activator, Vectored Thermal Pulse™ technology applies a combination of heat and pressure to the inner eyelid to safely remove gland obstructions and stagnant gland content. Therapeutic motion provides proximal-to-distal peristalsis to clear gland contents.
  Arms: Lipiflow - All Subjects
Device: iLux System — The iLux™ System is used to apply localized heat and pressure to a patient's eyelids. The system consists of a handheld instrument coupled to a single-use, sterile disposable component that is positioned to bridge the eyelid. The iLux device allows view of the eyelid through a magnifier, then warms the eyelid to 40 to 42˚C, then force-limited compression is applied manually to express the melted meibum from obstructed glands. Warming is accomplished using light energy emitted from LEDs in the Instrument. The LEDs are located behind a clear window on the open end of the Shroud. Two wavelengths of light are used: lime-green (568 nm) and near-infrared (850 nm). A mechanism in the Instrument allows the operator to apply pressure to the eyelid by controlling the movement of the Outer Pad using finger pressure applied to the Compression Control button. The force applied to the Compression Control is measured by a sensor in this mechanism.
  Arms: iLux - All Subjects

SUMMARY:
This study was designed to compare patient acceptance, comfort, and preference between two meibomian gland clearing devices (Lipiflow vs, iLux). Primary Objective was to compare patient comfort as assessed by Likert-style scale questionnaire following each bilateral procedure. Secondary Objective was to compare overall experience and treatment preference as assessed by Likert-style questionnaire following each bilateral procedure. Both devices are exempt from IDE regulations [21 CFR 812.2(c)].

DETAILED DESCRIPTION:
Introduction Meibomian gland disease (MGD) is increasingly recognized as a primary cause or contributor to tear instability and dry eye disease. Effective management of this disorder often requires meibomian gland expression and clearance. A variety of devices which apply pressure, heat or a combination of both to the glands have been used.

Two such devices that apply heat and pressure simultaneously are commercially available. LipiFlow (JNJ Vision Care) is an automated computer-controlled device that uses vectored thermal (hydraulic) pulsation applied by an activator device placed on the eye between the globe and the eyelids to achieve gland clearance. The iLux System (Alcon) is an operator controlled assisted manual device which applies heat generated by infrared LEDs and expression through cam driven mechanical pressure applied to the lids.

Device Descriptions LipiFlow Thermal Pulsation System

The Lipiflow Thermal Pulsation System is a commercially available device used in the treatment of MGD. It is cleared to be marketed by the United States Food and Drug Administration. The LipiFlow Thermal Pulsation System is intended for the application of localized heat and pressure therapy in adult patients with chronic cystic conditions of the eyelids, including meibomian gland dysfunction (MGD), also known as evaporative dry eye or lipid deficiency dry eye.

The LipiFlow Console provides the user interface and control elements of the system, including all software, algorithms and control elements. The Activator, a single-use sterile device, delivers automated therapeutic energies to each meibomian gland. Its contoured design vaults the cornea and protects the eye allowing a maximum therapeutic temperature of 43 degrees Celsius to reach glands from the inner eyelid, without damaging the eyelid or delicate structures of the globe. Insulation protects the cornea from exceeding a safe 39.5 degrees Celsius, while a pressure feedback loop sends pulsed sequences to expel blockages. Force equalization protects the globe from pressure transmission by focusing energy only on the eyelid. Delivered through the LipiFlow Activator, Vectored Thermal Pulse™ (VTP) technology applies a combination of heat and pressure to the inner eyelid to safely remove gland obstructions and stagnant gland content. Vectored heat and adaptive force equalization target the pulse, heat, and pressure on the meibomian glands to maximize effectiveness. Therapeutic motion provides proximal-to-distal peristalsis to clear gland contents.

iLux System

The iLux™ System is a medical device commercially available for use by Eye Care Professionals (ECP) to apply localized heat and pressure therapy to a patient's eyelids. It is cleared to be marketed by the United States Food and Drug Administration. The system consists of a handheld instrument coupled to a single-use, sterile disposable component that is positioned to bridge the eyelid. The iLux device allows an ECP to view the eyelid margin through a magnifier, then warm the eyelid tissue to a range of 40 to 42˚C, and then apply force-limited compression to the eyelid in order to express melted meibum from obstructed glands. The iLux System is indicated for the application of localized heat and pressure therapy in adult patients with chronic cystic conditions of the eyelids, including meibomian gland dysfunction (MGD), also known as evaporative dry eye.

The iLux Instrument is a handheld, electronic instrument used together with the iLux disposable to apply heating and pressure to the eyelid. The Instrument includes electronic circuits that read sensors in the Inner and Outer Eyelid Pads to measure temperatures representative of inner and outer eyelid temperature, respectively. Warming is accomplished using light energy emitted from LEDs in the Instrument. The LEDs are located behind a clear window on the open end of the Shroud. Two wavelengths of light are used: lime-green (568 nm) and near-infrared (850 nm). A mechanism in the Instrument allows the operator to apply pressure to the eyelid by controlling the movement of the Outer Pad using finger pressure applied to the Compression Control button. The force applied to the Compression Control is measured by a sensor in this mechanism. A graphic Screen displays information for operating the Instrument during a treatment.

Study Purpose / Objectives This study is designed to compare patient acceptance, comfort, and preference between two meibomian gland clearing devices. Both devices are exempt from IDE regulations [21 CFR 812.2(c)]. Primary Objective is to compare patient comfort as assessed by Likert-style scale questionnaire following each bilateral procedure. Secondary Objective is to compare overall experience and treatment preference as assessed by Likert-style questionnaire following each bilateral procedure.

Background "Comparison Between iLux™ and LipiFlow® in the Treatment of Meibomian Gland Dysfunction" listed on ClincalTrials.gov looked at a 4-week efficacy comparison between the two treatment devices. Pain and discomfort data were collected regarding the two procedures but was not analyzed for significance due to no pre-trial hypothesis. The raw data shows lower pain and discomfort scores immediately following the procedure for the Lipiflow as compared to iLux with similar pre-treatment and one-day post post-treatment scores (Thornhill 2019). There is currently no published research on the patient acceptance, comfort, and preference comparing any meibomian gland emptying devices.

ELIGIBILITY:
Inclusion Criteria:

1. Subject can be of any gender or race
2. Subject must be 18 years of age or older at the time of informed consent

2. Subject must be able to understand and must sign an Informed Consent that has been approved by an IRB 3. Subject must have confirmed diagnosis of Meibomian Gland Dysfunction 4. Subject must agree to not wear contact lenses the day of the Study visit

Exclusion Criteria:

1. History of intraocular or oculoplastic surgery within 6 months of Screening visit
2. History of ocular injury or trauma, chemical burns, or limbal stem cell deficiency within 3 months of the Screening visit
3. Active ocular infection or active ocular inflammation (including allergic conjunctivitis, vernal or giant papillary conjunctivitis) at time of Screening visit
4. History of ocular surface abnormality that may compromise corneal integrity
5. History of treatment with LipiFlow or iLux in either eye in the last 6 months
6. Allergy to topical proparacaine eye drops

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Procedure Comfort | 5 minutes
  Likert-scale questionnaire: 1=strongly disagree, 2=disagree, 3=Undecided, 4=Agree, 5=strongly agree - 1 Question

SECONDARY OUTCOMES:
Procedure Experience | 5 minutes
  Likert-scale questionnaire: 1=strongly disagree, 2=disagree, 3=Undecided, 4=Agree, 5=strongly agree - 4 Questions
Patient Preference | 5 minutes
  Questionnaire: Lipiflow, iLux, No Preference

CONTACTS AND LOCATIONS:
Overall Officials: Arthur B Epstein, OD, Principal Investigator — Ophthalmic Research Consultants of Arizona
Locations (1):
- Phoenix Eye Care, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- See also: Comparison Between iLux™ and LipiFlow® in the Treatment of Meibomian Gland Dysfunction — https://clinicaltrials.gov/ct2/show/NCT03055832

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT04454983/Prot_SAP_000.pdf